CLINICAL TRIAL: NCT04668690
Title: A Randomized, Open-label, Active Controlled, Multi-center Phase 3 Clinical Study to Compare the Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Injection With Chidamide in Patients With Relapsed/Refractory PTCL.
Brief Title: Clinical Study of Mitoxantrone Hydrochloride Liposome Injection vs. Chidamide in Patients With Relapsed/Refractory PTCL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-013
Record Dates: First submitted 2020-11-30; First posted 2020-12-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Mitoxantrone Hydrochloride Liposome Injection (Experimental): Patients with relapsed/refractory PTCL will receive Mitoxantrone Hydrochloride Liposome Injection every 28 days (a cycle) for a maximum of 8 cycles. The dose of Mitoxantrone Hydrochloride Liposome Injection is 20 mg/m2.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Active Comparator: Chidamide (Active Comparator): Patients with relapsed/refractory PTCL will receive Chidamide 30 mg p.o., twice per week until disease progression.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — Drug: Liposomal mitoxantrone hydrochloride (20 mg/m2) administered as an intravenous infusion on day 1 of each 28-day cycle.
  Other Names: HE071; Liposomal Mitoxantrone Hydrochloride Injection
  Arms: Experimental: Mitoxantrone Hydrochloride Liposome Injection
Drug: Chidamide — Drug: Chidamide tablet (30 mg) is given to the patients p.o. 30 minutes after breakfast, twice per week with 3-day intervals.
  Arms: Active Comparator: Chidamide

SUMMARY:
This is a randomized, open-label, active controlled, multi-center, phase 3 clinical study to compare the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection with Chidamide in patients with relapsed/refractory Peripheral T Cell Lymphoma (PTCL).

DETAILED DESCRIPTION:
This study is a randomized, open-label, positive control, multicenter, phase Ⅲ study to compare the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection with Chidamide in patients with relapsed/refractory Peripheral T Cell Lymphoma (PTCL). The eligible patients will be randomly assigned to the experimental and control groups in a 1:1 ratio. The patients in experimental group will receive Mitoxantrone Hydrochloride Liposome Injection (20 mg/m2) once every 28 days for a maximum of 6-8 cycles. Patients in the control group will be treated with Chidamide (30 mg) twice per week with 3-day intervals until disease progression. Patients in the control group who had confirmed disease progression will have the option to switch to the liposomal mitoxantrone hydrochloride treatment. Patients will receive treatment until the completion of 6-8 cycles of treatment (this applies only to the experiment group), disease progression, intolerable toxicity, death, loss to follow-up, withdrawal (patient's decision or investigator's decision), whichever comes first. All patients will have post-treatment follow-up for disease status until disease progression/recurrence, initiation of new antitumor therapy, or being lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18, ≤75 years, no gender limitation;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2;
4. Histopathologically confirmed Peripheral T -cell Lymphoma (PTCL) according to World Health Organization (WHO) criteria (version 2016), with the subtypes as follows:

   1. Peripheral T-cell lymphoma, unspecified (PTCL, NOS);
   2. Angioimmunoblastic T-cell lymphoma (AITL);
   3. ALK+ systematic anaplastic large T-cell lymphoma (ALCL, ALK+);
   4. ALK-systematic anaplastic large T-cell lymphoma (ALCL，ALK-);
   5. Extranobal NK/T cell lymphoma (nasal type) (NKTCL);
   6. Other subtypes of PTCL which are appropriate to be enrolled in the opinion of the investigator.
5. Patients have relapsed or are refractory to at least one line of prior systemic therapy (anthracycline-containing regimen) for PTCL. Relapse is defined as recurrence after CR or progress after PR; refractory refers to the efficacy of 2 cycles of treatment is PD, or the efficacy of 4 cycles of treatment is SD;
6. Subjects have at least one measurable lesion in accordance with the Lugano evaluation criteria (version 2014): the long axis of the lymph node shall be>1.5 cm, the long axis of the extranodal lesions shall be>1.0 cm.
7. Subjects must provide a written pathology/histological diagnosis report during the screening period and must agree to provide a tumor tissue section or tumor/lymph node tissue specimen to be sent to the central laboratory.
8. Life expectancy ≥ 12 weeks;
9. During the screening period, the patients should meet the following requirements and have not received infusion of cell growth factor, platelet and granulocyte within 7 days of the hematology test; 1) Absolute value of neutrophils ≥ 1.5 × 109/L; absolute value of neutrophil ≥ 1.0 × 109/L in patients with involvement of bone marrow; 2) Hemoglobin ≥ 90 g/L (no red cell infusion within 14 days), hemoglobin ≥ 75 g/L in patients with involvement of bone marrow; 3) Platelet ≥ 75 × 109/L in patients without involvement of bone marrow; platelet ≥ 50 × 109/L in patients with involvement of bone marrow; 4) Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (total bilirubin ≤ 3 × ULN if bilirubin level increase is caused by lymphoma invading the liver); 5) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; if the elevated level of AST or ALT is caused by liver involvement, both AST and ALT shall be ≤ 5 × ULN); 6) Creatinine < 1.5 × ULN.
10. Eligible fertile patients (male and female) must agree to use an effective method of contraception (hormonal or barrier or abstinence) with their partners from the study initiation until at least 7 months after the last treatment; women of childbearing potential must have a negative serum pregnancy test within 14 days prior to enrollment.

Exclusion Criteria (Limit: 15,000 characters)

1. Patients with leukemia type PTCL (adult T-cell leukemia/lymphoma, etc.), or in lymphoma leukemia stage (malignant cell proportion of > 20% in bone marrow examination); or with central nervous system (CNS) involvement, or with complicated of hemophagocytic syndrome.
2. History of allergy and contraindications to the same class and excipients of the experimental drug.;
3. Patients have one of the following conditions in the previous anti-tumor treatments:1) Patients received mitoxantrone or liposome mitoxantrone within 6 months;2) Patients who was treated with Chidamide and the efficacy was evaluated as PD; Patients who was treated with Chidamide within 6 months (if the patients have been treated with Chidamide for no more than 2 weeks, had no clear evidence of PD and no intolerable toxicity during the treatment period, and discontinued therapy for other reasons, may be considered with the investigator's consent);3) Those receiving treatment of Adriamycin or other anthracyclines previously, with the total cumulative dose of > 360 mg/m2 (other anthracycline drugs: 1 mg of epirubicin/pyramycin/daunorubicin is equivalent to 0.5 mg of doxorubicin, 1 mg of deoxydaunorubicin is equivalent to 2 mg of doxorubicin);4) Those received anti-tumor treatment, including cytotoxic chemotherapy, radiotherapy and targeted drug therapy within 4 weeks prior to the first use of the study drug, or immunomodulators (thalidomide, lenalidomide) within 3 weeks; or hormone or herbal therapy with lymphoma as indication within 2 weeks;
4. Participated in other clinical studies and received therapy within 4 weeks prior to the first administration of the study drug;
5. Those received allogeneic hematopoietic stem cell transplantation previously and autologous hematopoietic stem cell transplantation within 6 months;
6. Adverse reactions from the previous anti-tumor treatment have not yet recovered (>Grade 1 in NCI-CTCAE [Version 4.03], with the exception of hair loss and pigmentation);
7. Subjects with the impaired cardiac function or significant heart disease, including but not limited to:1) Myocardial infarction, congestive heart failure and viral myocarditis occurred 6 months before screening; heart disease with symptoms requiring treatment and intervention, such as unstable angina, arrhythmia, etc.;2) Congestive heart failure of ≥Grade 2 according to the New York Heart Association Classification;3) Cardiac ejection fraction less than 50% or less than the lower limit of the reference range of the laboratory examination used in the Research Center;4) Persistent myocardial disease;5) QTc > 450 milliseconds, or congenital long QT syndrome.
8. Patients with active infection, including hepatitis B (positive hepatitis B virus surface antigen and HBV-DNA titer higher than the upper limit of the reference range) and hepatitis C (positive hepatitis C virus RNA and HCV-RNA titer higher than the upper limit of the reference range);
9. History of severe autoimmune disease and immunodeficiency, including positive for human immunodeficiency virus (HIV); or other acquired or congenital immune deficiency diseases; or a history of organ transplantation;
10. Patients with other malignant tumors in the past five years (except the cured non-melanoma skin basal cell carcinoma and cervical carcinoma in situ);
11. Major surgery within 6 weeks prior to screening. or have a surgical schedule during the study period;
12. Patients have significant gastrointestinal disorders that may affect the ingestion, transportation, or absorption of the drug (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.) during the screening period;
13. Patients have uncontrolled hypertension (systolic pressure of 180 mmHg and/or diastolic pressure of 110 mmHg after treatment); or type 2 diabetes that cannot be controlled by oral hypoglycemic drugs or insulin therapy;
14. The patients had a history of active bleeding within the previous 3 months before the screening;
15. History of mental illness or history of drug abuse or dependence;
16. Pregnant or lactating women;
17. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by the IRC | Up to 48 months
  PFS (progression-free survival) assessed by the Independent Review Committee (IRC)

SECONDARY OUTCOMES:
PFS assessed by investigators | Up to 48 months
  PFS (progression-free survival) assessed by investigators
ORR | Up to 48 months
  Objective response rate
TTR | Up to 48 months
  Time to response
DoR | Up to 48 months
  Duration of response
DoRR | Up to 48 months
  Duration of response rate
CR | Up to 48 months
  Complete response rate
OS | Up to 48 months
  Overall survival
The incidence of AE and SAE | Up to 48 months
  To identify the incidence of AE and SAE, abnormalities in clinical laboratory assessments, ECGs, echocardiography, vital sign assessments, and physical exams

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China